CLINICAL TRIAL: NCT03511469
Title: Effects of Kontralateral Training in Patients With Bankart Lesion
Brief Title: Kontralateral Training in Patients With Bankart Lesion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Taha İbrahim Yıldız, Uzm. Fzt. Taha İbrahim Yıldız, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BK 1233412
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Strenght of Rotator Cuff Muscles
Keywords: Kontralateral Education, Bankart, Rehabilitation, Shoulder,
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized Control, Parallel Group Study
Who Masked: Outcomes Assessor
Masking Description: All assesment will be conducted with another therapist who is not aware of patient's treatment groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Patients in this group will only received standardized rehabilitation protochol after Bankart surgery
  Interventions: Other: Control Group
- Isokinetic Group (Experimental): Patients in this group will receive concentric training for rotator cuff muscles with isokinetic device in addition the the standart rehabilitation protocol.
  Interventions: Other: Isokinetic Group

INTERVENTIONS:
Other: Control Group — Control Group: Standart rehabilitation
  Arms: Control Group
Other: Isokinetic Group — Concentric group: Standart rehabilitation + isokinetic training
  Arms: Isokinetic Group

SUMMARY:
The rate of re-dislocation after arthroscopic bankart repair is up to 30%. The most important dynamic structure that prevents re-dislocation is the rotator cuff muscles. The aim of our study is to investigate the efficacy of contralateral training on patients with arthroscopic Bankart surgery. Patients with arthroscopic Bankart surgery will be included in the study. The patients will be randomly assigned into 3 groups and the first group will be the control group, the second group will be the concentric group and the third group will be the eccentric group. Standard rehabilitation program will be applied to all groups until 3 months after surgery. Between 2nd and 12nd weeks after surgery, concentric strengthening program will be applied to the rotator cuff muscles with isokinetic dynamometer to the 2nd group. In group 3, the eccentric strengthening program will be applied to the rotator sheath muscles with the same isokinetic dynamometer from the 2nd week until 12nd week .

The strength of the rotator sheath muscles will be measured in pre-op period, post-op week 12 and post-op month 6 with the isokinetic dynamometer in all patients. In addition, functional tests will be performed in pre-op period and post-op 6 months (Y balance test for upper extremity, Closed Kinetic Chain Upper Extremity Stability Test and Medicine Ball Throw Test).

DETAILED DESCRIPTION:
The return to sport after bankart surgery is very high. Yet, the rate of re-dislocation after arthroscopic bankart repair is up to 30%. The most important dynamic structure that prevents re-dislocation is the rotator cuff muscles. The aim of our study is to investigate the efficacy of contralateral training on patients with arthroscopic Bankart surgery. Patients with arthroscopic Bankart surgery will be included in the study. The patients will be randomly assigned into 3 groups and the first group will be the control group, the second group will be the concentric group and the third group will be the eccentric group. Standard rehabilitation program will be applied to all groups until 3 months after surgery. Between 2nd and 12nd weeks after surgery, concentric strengthening program will be applied to the rotator cuff muscles with isokinetic dynamometer to the 2nd group. In group 3, the eccentric strengthening program will be applied to the rotator sheath muscles with the same isokinetic dynamometer from the 2nd week until 12nd week .

The strength of the rotator sheath muscles will be measured in pre-op period, post-op week 12 and post-op month 6 with the isokinetic dynamometer in all patients. In addition, functional tests will be performed in pre-op period and post-op 6 months (Y balance test for upper extremity, Closed Kinetic Chain Upper Extremity Stability Test and Medicine Ball Throw Test).

ELIGIBILITY:
Inclusion Criteria:

* Having isolated arthroskopic bankart surgery
* Having <3 dislocation number
* Accepting to participate in the study
* Having rehabilitation in our clinic

Exclusion Criteria:

* Revision surgery
* Additional problem like bony bankart or laterjet surgery
* Having > 3 disloccation before surgery
* Refusing to participate in the study
* Not participating to the exercise program more then twice

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
İsokinetic assessment | six months
  Muscle strenhgt assesment on isokinetic dynamometer

SECONDARY OUTCOMES:
Funtional assesment | siz monyhs
  Sport-spesific Functional tests

CONTACTS AND LOCATIONS:
Overall Officials: Irem Duzgun, Prof., Study Director — Director of the study
Locations (1):
- Hacettepe Univercity, Faculty of Physical Theraphy and Rehablitation, Altındağ, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Tjong VK, Devitt BM, Murnaghan ML, Ogilvie-Harris DJ, Theodoropoulos JS. A Qualitative Investigation of Return to Sport After Arthroscopic Bankart Repair: Beyond Stability. Am J Sports Med. 2015 Aug;43(8):2005-11. doi: 10.1177/0363546515590222. Epub 2015 Jun 15. PMID 26078450
- [Background] Manca A, Dragone D, Dvir Z, Deriu F. Cross-education of muscular strength following unilateral resistance training: a meta-analysis. Eur J Appl Physiol. 2017 Nov;117(11):2335-2354. doi: 10.1007/s00421-017-3720-z. Epub 2017 Sep 21. PMID 28936703